CLINICAL TRIAL: NCT00833001
Title: A Prospective, Multi-center Study to Evaluate the Clinical Performance of the GYNECARE PROLIFT + M* Pelvic Floor Repair System as a Device for Pelvic Organ Prolapse
Brief Title: Clinical Performance of the GYNECARE PROLIFT + M* Pelvic Floor Repair System as a Device for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 300-07-006
Record Dates: First submitted 2009-01-26; First posted 2009-01-30 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Cystocele; Rectocele; Enterocele
Keywords: Anterior vaginal prolapse (medial, lateral,apical cystocele); Posterior vaginal prolapse (rectocele and/or enterocele); Vault prolapse (enterocele, uterine/vaginal vault prolapse)
MeSH Terms: conditions — Cystocele; Rectocele; Hernia; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: GYNECARE PROLIFT+M* Pelvic Floor Repair System
  Interventions: Device: GYNECARE PROLIFT+M* Pelvic Floor Repair System

INTERVENTIONS:
Device: GYNECARE PROLIFT+M* Pelvic Floor Repair System — Pre-shaped mesh implants made of GYNECARE GYNEMESH M composite mesh, comprised of absorbable polyglecaprone 25 monofilament fiber and nonabsorbable polypropylene monofilament fiber
  Other Names: ULTRAPRO* mesh

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the PROLIFT system with a new lighter-weight mesh in repair of vaginal prolapse.

DETAILED DESCRIPTION:
Vaginal prolapse (a feeling of bulge in the vagina) may cause some distressing symptoms such as loss of control of the bowel or bladder, and may also cause problems with women's sex life. There are a number of different surgical procedures which are used to repair prolapse. Sometimes a mesh is placed in the pelvis to support the weakened tissues. There is a lot of research going on to find the most suitable type of mesh to repair vaginal prolapse. The GYNECARE PROLIFT + M* Pelvic Floor Repair system is similar to a mesh already used for this procedure called ULTRAPRO*, but is lighter in weight. Currently, ULTRAPRO* is only approved for use in hernia repair and is not licensed for gynecological procedures. This study will be the first clinical investigation of this mesh in vaginal prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic pelvic organ prolapse of ICS POP-Q Stage III or IV, suitable for surgical repair. Perineal repair, vaginal hysterectomy and/or mid urethral sling procedures for incontinence may be performed concurrently.
* Age > or = 18 years.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires, and documents this agreement by signing the Ethics Committee / IRB approved informed consent.

Exclusion Criteria:

* Additional surgical intervention for POP repair concurrent to the Gynecare Prolift+M procedure (e.g. paravaginal repair, sacrocolpopexy, colporrhaphy in a non-Gynecare Prolift+M treated compartment).
* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Previous hysterectomy within 6 months of scheduled surgery.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of any pelvic radiation therapy.
* History of chemotherapy within 6 months of the planned procedure.
* Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spina bifida, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 with symptomatic pelvic organ prolapse of ICS POP-Q Stage III or IV, suitable for surgical repair.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) score | 12 months post-procedure

SECONDARY OUTCOMES:
Summary of treated compartment ICS POP-Q stage | 3, 12, 24 and 36 months
Proportion of subjects with the leading edge within the hymen and without further re-intervention for POP | 12, 24 and 36 months
Incidence of de novo prolapse (a post-operative prolapse)only in the untreated compartment, provided there was no pre-operative defect in that compartment | Procedure to 36 months
Mean scores and change from baseline in PFDI-20 scores, including sub scores (POPDI, CRADI and UDI | 3, 12, 24 and 36 months
Mean scores and change from baseline in PFIQ-7, including sub-scores (POPIQ, CRAIQ and UIQ). | 3, 12, 24 and 36 months
Days to return to normal activities (walking, driving, work, household activities and sexual intercourse) | 1, 3, and 12 months
Assessment of sexual function using PISQ-12 (mean scores and change from baseline) in subjects sexually active at baseline | 12, 24 and 36 months
Incidence of new onset dyspareunia, resolution or continuance of pre-existing dyspareunia | Baseline to 36 months
Adverse Events | Procedure to 36 months
Determination of any exposures/erosions including location | Procedure to 36 months
Summary of International Continence Society (ICS) Stages | 3, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (8):
- Sint Lodewijkstraat 78, Genk, Belgium
- CHRU de Lille, Lille, France
- Germany (5):
  - DRT Krankenhaus, Chemnitz
  - Martin Luther University, Halle
  - Kreiskrankenhaus, Hamelin
  - Universitatsklinik Tubingen, Tübingen
  - St. Marien-Hospital, Vechta
- Reinier de Graaf Gasthuis, Delft, Netherlands

REFERENCES:
- [Result] Milani AL, Hinoul P, Gauld JM, Sikirica V, van Drie D, Cosson M; Prolift+M Investigators. Trocar-guided mesh repair of vaginal prolapse using partially absorbable mesh: 1 year outcomes. Am J Obstet Gynecol. 2011 Jan;204(1):74.e1-8. doi: 10.1016/j.ajog.2010.08.036. Epub 2010 Oct 20. PMID 20965491